CLINICAL TRIAL: NCT01571570
Title: A Phase I, Open-Label, Randomized, 3-Panel, 3-way Crossover Trial in Healthy Adult Subjects to Assess the Relative Bioavailability of TMC435 Following Administration of 2 Liquid Formulations or 2 Different Capsule Concept Formulations Compared ot the Phase III 150 mg Capsule, and to Assess the Effect of Food on the Bioavailability of TMC435 Following Administration of the Liquid Formulations.
Brief Title: A Study to Assess Bioavailability & Food Effect of Different Liquid and Capsule Formulations of TMC435.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen R&D Ireland (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR100787; TMC435HPC1002 (Other: Janssen R&D Ireland)
Record Dates: First submitted 2012-01-23; First posted 2012-04-05 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Healthy Volunteers
Keywords: Healthy volunteers; Food effect; Capsule; Formulations; Liquid formulation; Concept K; Concept L; Oral suspension; Oral solution; TMC435HPC1002; TMC435; HPC
MeSH Terms: interventions — Simeprevir; Suspensions; Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (9):
- Treatment A (Experimental): Panel 1: single oral dose of 150 mg TMC435 150 mg capsule, fed
  Interventions: Drug: TMC435 150 mg capsule
- Treatment B (Experimental): Panel 1: single oral dose of 150 mg TMC435 oral suspension (20 mg/mL), fasted
  Interventions: Drug: TMC435 150 mg oral suspension (20 mg/mL)
- Treatment C (Experimental): Panel 1: single oral dose of 150 mg TMC435 oral suspension (20 mg/mL), fed
  Interventions: Drug: TMC435 150 mg oral suspension (20 mg/mL)
- Treatment D (Experimental): Panel 2: single oral dose of 150 mg TMC435 150 mg capsule, fed
  Interventions: Drug: TMC435 150 mg capsule
- Treatment E (Experimental): Panel 2: single oral dose of 150 mg TMC435 oral solution (10 mg/mL), fasted
  Interventions: Drug: TMC435 150 mg oral solution (10 mg/mL)
- Treatment F (Experimental): Panel 2: single oral dose of 150 mg TMC435 oral solution (10 mg/mL), fed
  Interventions: Drug: TMC435 150 mg oral solution (10 mg/mL)
- Treatment G (Experimental): Panel 3: single oral dose of 150 mg TMC435 150 mg capsule, fed
  Interventions: Drug: TMC435 150 mg capsule
- Treatment H (Experimental): Panel 3: single oral dose of 150 mg TMC435 capsule concept K, fed
  Interventions: Drug: TMC435 150 mg capsule concept K
- Treatment I (Experimental): Panel 3: single oral dose of 150 mg TMC435 capsule concept L, fed
  Interventions: Drug: TMC435 150 mg capsule concept L

INTERVENTIONS:
Drug: TMC435 150 mg capsule — single oral dose of 150 mg TMC435 150 mg capsule
  Other Names: TMC435
  Arms: Treatment A; Treatment D; Treatment G
Drug: TMC435 150 mg oral suspension (20 mg/mL) — single oral dose of 150 mg TMC435 oral suspension
  Other Names: TMC435
  Arms: Treatment B; Treatment C
Drug: TMC435 150 mg oral solution (10 mg/mL) — single oral dose of 150 mg TMC435 oral solution
  Other Names: TMC435
  Arms: Treatment E; Treatment F
Drug: TMC435 150 mg capsule concept K — single oral dose of 150 mg TMC435 capsule concept K
  Other Names: TMC435
  Arms: Treatment H
Drug: TMC435 150 mg capsule concept L — single oral dose of 150 mg TMC435 capsule concept L
  Other Names: TMC435
  Arms: Treatment I

SUMMARY:
The purpose of this study is to evaluate the relative bioavailability and the short-term safety and tolerability of TMC435 following administration of 3 single oral doses of 150 mg, given as different formulations in healthy adult participants. In addition, this study is to assess for the acceptability of the taste of both liquid formulations.

DETAILED DESCRIPTION:
TMC435 is being investigated for the treatment of chronic hepatitis C infection. The current study is a Phase I, open-label (both participant and investigator know the name of the medication given at certain moment), randomized (study medication is assigned by chance) study designed to assess the relative bioavailability and food effect of 2 liquid formulations of TMC435, currently being developed for potential pediatric use, compared to the Phase III 150 mg capsule. Also new capsule concept formulations will be investigated in comparison with the Phase III 150 mg capsule. The study will be performed in healthy adult participants and is divided over 3 panels. Participants will be randomized within a panel. Each participant will receive 3 different treatments according to a classical 6-sequence, 3-period Williams design. In Panel 1 and Panel 2, a single oral dose of 150 mg TMC435 oral suspension respectively with other strength will be compared with the capsule used in Phase III. In Panel 3, two different capsule concept formulations will be compared with the capsule used in Phase III. In panels containing the liquids, formulations will be compared under fasted and fed conditions to investigate the food effect. In all treatments, the participants will receive medication on Day 1 of each treatment. There will be a washout period of at least 7 days between subsequent treatments. The main focus of the trial is the pharmacokinetic characteristics of all formulations (level-profile of TMC435 over time in the blood stream). This evaluation requires multiple blood samples from Day 1 till Day 4 in each treatment. Safety assessments (blood and urine tests, blood pressure, pulse, electrocardiogram, and physical examination) will follow a different schedule and will be evaluated from signing of the Informed Consent Form onwards until the last trial-related visit throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers should be healthy on the basis of physical examination, medical history, laboratory tests, 12-lead electrocardiogram and vital signs, performed at screening, have a body Mass Index (BMI, weight in kg divided by the square of height in meters) of 18.0 to 30.0 kg/m2, extremes included and be non-smoking for at least 3 months prior to screening.
* Women must be postmenopausal for at least 2 years and/or surgically sterile or not heterosexually active for duration of the trial.

Exclusion Criteria:

* All participants with known allergies, hypersensitivity or intolerance to TMC435 or any of the excipients.
* Use of concomitant medication, including over the counter products, herbal medication and dietary supplements, except for paracetamol (acetaminophen) or ibuprofen.
* Any condition that, in the opinion of the investigator, would compromise the study or well-being of the participant or prevent the subject from meeting or performing study requirements.
* History or suspicion of current use of alcohol, barbiturate, amphetamine, recreational or narcotic drug use, which in investigator's opinion would compromise participant's safety and/or compliance with the trial procedures.
* Participation in an investigational drug trial with TMC435.
* Infected with HIV or Hepatitic A, B or C.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2012-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Comparing the bioavailability of oral solution and oral suspension formulation with the capsule formulation of TMC435 (fed state) | 4 days
  Comparing the rate and extent of absorption (bioavailability) of 2 different liquid formulations (oral suspension [150 mg ie, 20 mg/mL] and oral solution [150 mg ie, 10 mg/mL]) versus capsule formulation (150 mg) of TMC435, after a high-fat breakfast (fed state)
Comparing the bioavailability of oral solution and oral suspension formulation of TMC435 in fed and fasted state | 4 days
  Comparing the rate and extent of absorption (bioavailability) of 2 different liquid formulations (oral suspension [150 mg ie, 20 mg/mL] and oral solution [150 mg ie, 10 mg/mL]) of TMC435 in fed state (high-fat breakfast) versus fasted state
Comparing the bioavailability of concept K capsule and concept L capsule formulation with the capsule formulation of TMC435 (fed state) | 4 days
  Comparing the rate and extent of absorption (bioavailability) of 2 different capsule formulations (concept K capsule [150 mg] and concept L capsule [150 mg]) versus capsule formulation (150 mg) of TMC435 after a high-fat breakfast (fed state)

SECONDARY OUTCOMES:
Number of participants with adverse events | 18 days
  Adverse events, abnormal clinical laboratory findings, abnormalities assessed in vital signs examination, physical examination, ECG measurements were evaluated for safety and tolerability during the study
Acceptability of taste assessed by taste questionnaires | Day 1 of Treatment B and E
  Taste Questionnaires used to assess taste acceptability of oral suspension and solution of TMC435 under fasted conditions. Taste Questionnaire for adults: participant had to select appropriate choice (None, Weak, Moderate, Strong) for 3 different types of tastes "Sweetness, Bitterness, Flavour" and also select appropriate choice (Bad, Amost acceptable, Acceptable and Good) for the Overall taste. For pediatric participants: fill the visual analog scale by selecting appropriate choice (Dislike it very much, Dislike it a little, Not sure, Like it a little and Like it very much)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen R&D Ireland Clinical Trial, Study Director — Janssen R&D Ireland
Locations (1):
- Harrow, United Kingdom